CLINICAL TRIAL: NCT01427985
Title: The Influence of Two Different Premedication Protocols for Endotracheal Intubation in Neonates on Cerebral Oxygenation
Brief Title: Influence of Premedication Protocols for Neonatal Endotracheal Intubation on Cerebral Oxygenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manuel Schmid, Dr. med., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULMNEONIRS02
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Newborn; Preterm; Intubation
MeSH Terms: conditions — Premature Birth | interventions — Atropine; Fentanyl; Mivacurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation followed by analgosedation (Experimental): Give Atropin, then Mivacurium, immediately followed by Fentanyl
  Interventions: Drug: Atropine, Fentanyl, Mivacurium
- Analgosedation followed by Relaxation (Active Comparator): Give atropin, then Fentanyl, then Mivacurium
  Interventions: Drug: Atropine, Fentanyl, Mivacurium

INTERVENTIONS:
Drug: Atropine, Fentanyl, Mivacurium — 1. Atropin 10µg/kg
  2. Mivacurium 200µg/kg immediately followed by
  3. Fentanyl 2µg/kg
  Arms: Relaxation followed by analgosedation
Drug: Atropine, Fentanyl, Mivacurium — 1. Atropin 10µg/kg
  2. Fentanyl 2µg/kg, repeat max. two times
  3. Mivacurium 200µg/kg
  Arms: Analgosedation followed by Relaxation

SUMMARY:
The purpose of this study is to examine the influence of premedication drugs Atropin, Fentanyl and Mivacurium and of endotracheal intubation on cerebral oxygenation and cardiac output in term and preterm newborn infants. Two different protocols of premedication are compared.

DETAILED DESCRIPTION:
Influence of the following procedures will be examined:

* Application of Atropin
* Application of Fentanyl
* Application of Mivacurium
* possible desaturation and / or bradycardia during intubation attempts
* restoration of arterial oxygen saturation and / or heart rate after succesful intubation

We aim to examine the change of the following parameters by the use of electrical cardiometry:

* stroke volume
* cardiac output

We compare two different premedication protocols and we evaluate the impact of these protocol on the time needed for intubation and on intubation difficulties .

ELIGIBILITY:
Inclusion Criteria:

* newborn infant below 44 weeks postmenstrual age
* indication for elective or semi-elective endotracheal Intubation
* parental informed consent

Exclusion Criteria:

* emergency intubation

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change of cerebral tissue oxygen saturation during premedication and intubation | from 1 minute before first study drug until 10 minutes after end of procedure
  A baseline value of cerebral tissue oxygen saturation before first application of premedication drugs is determined. Change of cerebral tissue oxygen saturation is defined as area under this threshold from first drug application until recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel B Schmid, Dr. med., Principal Investigator — University of Ulm
Locations (1):
- University Medical Center, Ulm, Baden-Wurttemberg, Germany